CLINICAL TRIAL: NCT05985707
Title: The Efficacy and Safety of KN026 Combination Chemotherapy ± KN046 in HER2-Positive Advanced Colorectal Cancer and Biliary Tract Cancer as First-Line Treatment： a Phase Ⅱ Study
Brief Title: KN026 Plus Chemotherapy ± KN-046 in HER2 Positive Colorectal Cancer and Biliary Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HERCKER-01
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: HER2-positive Colorectal Cancer; HER2-positive Biliary Tract Cancer
MeSH Terms: interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Experimental): Arm A will include HER2-positive treatment-naive metastatic colorectal cancer patients, and the patients in this cohort will receive XELOX and KN026 treatment.
  Interventions: Drug: KN026; Drug: XELOX
- B (Experimental): Arm B will include HER2-positive treatment-naive metastatic colorectal cancer patients, and the patients in this cohort will receive XELOX and KN026 + KN046 treatment.
  Interventions: Drug: KN026; Drug: KN046; Drug: XELOX
- C (Experimental): Arm C will include HER2-positive treatment-naive metastatic biliary tract cancer patients, and the patients in this cohort will receive XELOX and KN026 + KN046 treatment.
  Interventions: Drug: KN026; Drug: KN046; Drug: XELOX

INTERVENTIONS:
Drug: KN026 — KN026 is a novel bispecific antibody that simultaneously binds to two distinct HER2 epitopes.
Drug: KN046 — KN046 is a novel bispecific antibody that blocks both PD-L1 interaction with PD-1 and CTLA-4 interaction with CD80/CD86.
  Arms: B; C
Drug: XELOX — XELOX is the standard first-line chemotherapy in metastatic colorectal cancer and biliary duct cancer.

SUMMARY:
The goal of this Interventional clinical trial is to learn about the efficacy and safety of KN026 and chemotherapy ± KN046 in HER2-positive metastatic colorectal cancer and biliary tract cancer. Participants will receive standard first-line chemotherapy (capecitabine + oxaliplatin) combined with KN026 (a HER2-targeted bispecific antibody) ± KN046 （a PD-L1/CTLA-4 targeted bispecific antibody）.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are able to comprehend the informed consent information and sign the informed consent form.
2. Participants ≥ 18 years old, of any gender.
3. Cohorts A and B: Histologically confirmed unresectable HER2-positive metastatic colorectal cancer, meeting the following criteria: a) Previously untreated with systemic anti-tumor therapy, or the time from (neo)adjuvant chemotherapy completion to disease recurrence > 6 months; b) Gene sequencing shows wild-type RAS and BRAF (participants' previous KRAS and BRAF test results are acceptable).
4. Cohort C: Histologically confirmed unresectable HER2-positive biliary tract cancer, including intrahepatic or extrahepatic bile duct cancer or gallbladder cancer: a) Previously untreated with systemic anti-tumor therapy; b) If previously received (neo)adjuvant radiotherapy, the time from treatment completion to disease recurrence is > 6 months.
5. HER-2 positive defined as a) HER2 IHC 3+; b) HER2 IHC 2+ with HER2 amplification (HER2/CEP17 > 2.0 by ISH method)； c) HER copy number > 6 by next-generation sequencing using tumor tissue or circulating tumor DNA.
6. LVEF ≥ 50%

(9) Within 7 days before the first administration, hepatic function should meet the following criteria:

* Total bilirubin ≤ 1.0 x ULN (≤ 1.5 x ULN for subjects with Gilbert's syndrome or liver metastases)
* Transaminases (ALT/AST) ≤ 1.5 x ULN (≤ 3 x ULN for subjects with liver metastases) (10) Within 7 days before the first administration, renal function should be as follows:
* Serum creatinine ≤ 1.5 x ULN
* Creatinine clearance ≥ 60 mL/min (calculated using the Cockcroft-Gault formula) (11) Within 7 days before the first administration, bone marrow function should meet the following criteria:
* Hemoglobin ≥ 90 g/L
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L (12) TSH within the normal range; if TSH is abnormal, free T3 and free T4 should be within the normal range.

  (13) Expected survival of ≥ 3 months. (14) Participants need to receive capecitabine and oxaliplatin regimen chemotherapy based on clinical assessment.

  (15) Female participants of childbearing potential or male participants with partners of childbearing potential must agree to use effective contraception from 7 days before the first dose until 24 weeks after the last dose. Female participants of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose.

  (16) Participants are capable and willing to comply with the study protocol, treatment plan, laboratory tests, and other study-related procedures.

Exclusion Criteria:

1. Subjects with untreated active brain metastases or leptomeningeal metastases; if subjects have received treatment for brain metastases and the lesions are stable (stable brain imaging for at least 4 weeks before the first dose with no evidence of new or enlarging brain lesions and no new neurological symptoms or stable neurological symptoms at baseline), they are allowed to be enrolled.
2. Ampullary carcinoma.
3. Previous history of receiving any systemic anticancer therapy for metastatic tumors or participation in interventional clinical trials.
4. Within 14 days before the first dose, the subject requires a continuous 7-day treatment of systemic corticosteroids (≥10 mg/day prednisone or equivalent of other corticosteroids) or immunosuppressive agents; exceptions are inhaled or locally applied corticosteroids or physiological replacement doses of corticosteroids for adrenal insufficiency. Short-term (≤7 days) corticosteroids are allowed for prevention (e.g., contrast dye allergy) or treatment of non-autoimmune conditions (e.g., delayed hypersensitivity reactions caused by exposure to allergens).
5. Received live vaccines (including attenuated live vaccines) within 28 days before the first dose.
6. Subjects with interstitial lung disease or requiring oral or intravenous administration of corticosteroids.
7. History or current presence of autoimmune diseases, including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener's granulomatosis (granulomatosis with polyangiitis), Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, autoimmune hepatitis, systemic sclerosis (scleroderma), Hashimoto's thyroiditis (except under certain circumstances as outlined below), autoimmune vasculitis, and autoimmune neurological disorders (such as Guillain-Barre syndrome). The following conditions are exempted: type 1 diabetes, stable hypothyroidism on hormone replacement therapy (including hypothyroidism caused by autoimmune thyroid disease), and psoriasis or vitiligo not requiring systemic treatment.
8. History of another malignant tumor within 5 years before the first dose, except for cured skin squamous cell carcinoma, basal cell carcinoma, non-muscle-invasive bladder cancer, localized low-risk prostate cancer (defined as stage ≤T2a, Gleason score ≤6, and prostate-specific antigen (PSA) ≤10 ng/mL at diagnosis, and patients who received curative treatment without PSA biochemical recurrence), and in situ cervical/breast cancer.
9. Has uncontrolled comorbidities, including but not limited to the following conditions:

   * Active HBV or HCV infection.
   * Subjects with positive HBsAg and/or HCV antibodies during screening must undergo HBV DNA and/or HCV RNA testing. Subjects with HBV DNA ≤ 500 IU/mL (or ≤ 2000 copies/mL) and/or HCV RNA negative can be enrolled; during the trial, the investigator will decide on monitoring HBV DNA based on the subject's situation.
   * Known HIV infection or history of AIDS.
   * Active tuberculosis.
   * Active infection or systemic use of antimicrobial drugs for more than 1 week within 28 days before the first dose of this study; unexplained fever within 2 weeks before dosing.
   * Uncontrolled hypertension (resting blood pressure ≥ 160/100 mmHg), symptomatic heart failure (NYHA class II-IV), unstable angina or myocardial infarction within the past 6 months, or risk of QTc prolongation or arrhythmia (baseline QTc > 470 msec corrected by Fridericia method, difficult-to-correct hypokalemia, long QT syndrome, resting heart rate > 100 bpm with atrial fibrillation, or severe valvular heart disease).
   * Active bleeding that cannot be controlled even with medical intervention.
10. History of allogeneic bone marrow or organ transplantation.
11. History of allergic reactions, hypersensitivity, or intolerance to antibody-based drugs; history of significant drug allergies (e.g., severe allergic reactions, immune-mediated hepatotoxicity, immune-mediated thrombocytopenia, or anemia).
12. Pregnant and/or lactating females.
13. Other conditions that, in the opinion of the investigator, may affect the safety or compliance of the study drug treatment, including but not limited to moderate to large pleural/peritoneal/pericardial effusion, difficult-to-correct pleural/peritoneal/pericardial effusion, intestinal obstruction or subacute intestinal obstruction, psychiatric disorders, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Objective response rate (defined as CR+PR) is reported based on investigator's evaluation.

SECONDARY OUTCOMES:
Progression free survival | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Progression-free survival (PFS) is defined as the time from the date of the first dose to the earlier of the dates of the first objective documentation of radiographic progressive disease (PD) or death due to any cause.
Duration of response | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Duration of response (DOR) is defined as the time from the date of the first response to the first objective documentation of radiographic progressive disease (PD) or death due to any cause.
Disease control rate | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Disease control rate (defined as CR+PR+SD) is reported based on investigator's evaluation.
Time to response | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Time to response (TOR) is defined as the time from the date of the first dose to the first objective documentation of radiographic objective response.
Overall survival | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Overall survival (OS) is defined as the time from the date of first dose to the date of death from any cause.
Frequency of adverse events | From the date of signing the informed consent form up to 30 (+7) days after last dose.
  A treatment-emergent adverse event (TEAE) is defined as any adverse event not present prior to the initiation of drug treatment or any adverse event already present that worsens in intensity or frequency following exposure to the drug treatment. TEAEs were graded using National Cancer Institute (NCI)-CTCAE version 4.03.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University cancer hospital & institution, Beijing, State*, China

IPD SHARING:
Plan to Share IPD: No